CLINICAL TRIAL: NCT01831661
Title: A Randomized, Open Label, Two-treatment, Two -Period, Two-sequence, Single Dose, Crossover, Oral Bioequivalence Study of Metformin Hydrochloride Extended-Release Tablets USP 750 mg of Ipca Laboratories Ltd, India and GLUCOPHAGE®XR (Metformin HCl Extended-release Tablets) 750 mg of Bristol-Myers Squibb Company, USA in Normal, Healthy, Adult, Human Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Metformin Hydrochloride Extended-Release Tablets USP 750 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IPCA Laboratories Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-VIN-183
Record Dates: First submitted 2013-04-06; First posted 2013-04-15 (Estimated); Last update posted 2013-04-15 (Estimated); Status verified 2013-04

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GLUCOPHAGE®XR (Active Comparator): GLUCOPHAGE®XR (Metformin HCl extended-release tablets) 750 mg of Bristol-Myers Squibb Company, USA
  Interventions: Drug: Metformin Hydrochloride Extended-Release Tablets USP 750 mg; Drug: GLUCOPHAGE®XR
- Metformin Hydrochloride Extended-Release Tablets USP 750 mg (Experimental): Metformin Hydrochloride Extended-Release Tablets USP 750 mg of Ipca Laboratories Ltd, India
  Interventions: Drug: Metformin Hydrochloride Extended-Release Tablets USP 750 mg; Drug: GLUCOPHAGE®XR

INTERVENTIONS:
Drug: Metformin Hydrochloride Extended-Release Tablets USP 750 mg — Metformin Hydrochloride Extended-Release Tablets 750 mg once a day
  Other Names: Test Product
Drug: GLUCOPHAGE®XR — GLUCOPHAGE®XR 750 mg once a day
  Other Names: Reference product

SUMMARY:
The study was a randomized, open label, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study in normal, healthy adult human subjects under fasting condition.

DETAILED DESCRIPTION:
Objective of the study is to compare and evaluate the single-dose oral bioavailability of Metformin Hydrochloride Extended-Release Tablets USP 750 mg of Ipca Laboratories Ltd, India and GLUCOPHAGE®XR (Metformin HCl extended-release tablets) 750 mg of Bristol-Myers Squibb Company, USA in normal, healthy, adult, human subjects under fasting condition.

Total duration of the study was of 17 days from the day of admission of first period till the end of second period.

Upon entering into the study, subjects were housed in clinical facility of Veeda Clinical Research Pvt. Ltd. to ensure 10 hours overnight fasting before dosing and continued to be housed in the facility till 36.00 hours post-dose blood sample collection in each of the two periods.

A gap of 14 days was kept as wash out between each consecutive dosing period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged between 18 and 45 years (including both).
2. Subjects' weight within normal range according to normal values for Body Mass Index (18.5 to 24.9 kg/m2) (including both) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within clinically acceptable normal range.
4. Subjects having clinically acceptable 12-lead electrocardiogram (ECG).
5. Subjects having clinically acceptable chest X-Ray (PA view).
6. Subjects having negative urine screen for drugs of abuse (including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Subjects having negative alcohol breathe test.
8. Subjects willing to adhere to protocol requirements and to provide written informed consent.
9. Subjects having negative Beta-hCG Pregnancy test (only for female subjects).
10. For Female Subjects:

1) Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies, diaphragm, intrauterine device (IUD), or abstinence, or 2) Postmenopausal for at least 1 year, or if less than 1 year, then following acceptable contraceptive measures as mentioned above 3) Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject).

Exclusion Criteria:

1. Hypersensitivity to Metformin or to any excipients or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological, neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting
4. History or Presence of significant alcoholism or drug abuse.
5. History or presence of significant asthma, urticaria or other allergic reactions.
6. History or presence of significant gastric and/or duodenal ulceration.
7. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
8. History or presence of cancer.
9. History or presence of significant easy bruising or bleeding.
10. History or presence of significant recent trauma.
11. Subjects who have been on an abnormal diet (for whatever reason) during four weeks preceding the study.
12. Difficulty with donating blood.
13. Difficulty in swallowing solids like tablets or capsules.
14. Use of any prescribed or OTC medication during last two weeks prior to dosing in period 01.
15. Consumption of grapefruit juice, xanthine-containing products, tobacco containing products or alcohol within 48 hours prior to dosing.
16. Major illness during 3 months before screening.
17. Participation in a drug research study within past 3 months.
18. Donation of blood from past 3 months before screening.
19. Female subjects who are currently breast feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters. | 1 Months
  Pre-dose & at 1.00, 2.00, 3.00, 4.00, 4.50, 5.00, 5.50, 6.00, 6.50, 7.00, 8.00, 9.00, 10.00, 12.00, 16.00, 20.00, 24.00, 30.00 and 36.00 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Hardik Dave, M.B.B.S, Principal Investigator — Veeda Clinical Research Pvt. Ltd.
Locations (1):
- Veeda Clinical Research Pvt. Ltd., Ahmedabad, Gujarat, India